CLINICAL TRIAL: NCT01672346
Title: Pulmonary Vein (PV) Reconnection After Pulmonary Vein Antrm Isolation (PVAI) at Different Power Settings and Adenosine Provocation
Brief Title: PV Reconnection After PVAI at Different Power Settings and Adenosine Provocation
Acronym: ZODIAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: California Pacific Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive medical director, TCAI, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZODIAC_TCAI
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: PAF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): PVAI with ablation of posterior wall contained within pulmonary veins using energy up to 30 watts and post-ablation adenosine challenge
  Interventions: Procedure: PVAI followed by adenosine provocation
- Arm II (Active Comparator): AF ablationPVAI with ablation of posterior wall contained within pulmonary veins using energy up to 40 watts and post-ablation adenosine challenge
  Interventions: Procedure: PVAI followed by adenosine provocation

INTERVENTIONS:
Procedure: PVAI followed by adenosine provocation — All patients will undergo PVAI and ablation of the posterior wall of the LA using an open-irrigated ablation catheter and under general anesthesia. After PV isolation is achieved, all will undergo PVAI followed by adenosine provocation test with 24 mg of adenosine to check for PV reconnection. Upon identification, additional RF energy would be used to ablate those sites (that were revealed by adenosine-provocation).

SUMMARY:
In this prospective randomized study, we aim to compare the rate of PV reconnection following PVAI performed at different energy settings (30 Watts vs 40 Watts) where dormant PV conduction will be unmasked by adenosine-provocation.

DETAILED DESCRIPTION:
Background:

The efficiency of catheter ablation in drug-refractory atrial fibrillation (AF) is compromised by high incidence of post-ablation AF recurrences requiring multiple ablation procedures (1). Post-PVAI (pulmonary vein antrum isolation) AF recurrence is mostly due to reconnection of the previously isolated PVs (2). Earlier studies have revealed that elimination of dormant PV conduction revealed by adenosine-provocation ensures better outcome as reconnection mostly happens due to presence of incompletely ablated tissue and identification and complete ablation decrease chance of recurrence (1). Adenosine is specifically chosen for induction of triggers because it is known to transiently or permanently re-establish left atrium-pulmonary vein (LA-PV) conduction after apparently successful PV isolation (3). Datino et al have demonstrated in the canines that adenosine selectively hyperpolarizes the PVs by increasing inward rectifier potassium (K+) current and restores excitability (4). As incompletely ablated tissue can potentially cause AF recurrence, the depth and extension of the lesion are crucial factors in determining the success-rate of ablation; these in turn are directly influenced by catheter type and the radio-frequency (RF) energy settings (5). In a previous study, Matiello et al have reported cooled-tip catheter at 40w setting to be more effective in preventing recurrence than that with 30w setting (5). However, none of the earlier studies have examined the rate of PV reconnection when AF ablation is done at different power settings using open-irrigated catheters after the dormant sites are revealed by adenosine-challenge.

Hypothesis:

Use of higher wattage during ablation before and after adenosine-challenge is associated with lower rate of PV reconnection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients presenting with drug-refractory PAF undergoing first ablation
3. Ability to understand and provide signed informed consent

Exclusion Criteria:

1. Previous catheter ablation or MAZE procedure in left atrium
2. Reversible causes of atrial arrhythmia such as hyperthyroidism, sarcoidosis, pulmonary embolism etc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2013-05; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | 1 year
  Recurrence of AF due to PV reconnection AF recurrence is defined as any episode of AF/AT (atrial tachycardia) longer than 30 seconds will be considered as recurrence. Episodes that occur during the first 3 months of the procedure (blanking period) will not be considered as recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — TCAI
Locations (2):
- United States (2):
  - St. david's Medical Center, Austin, Texas
  - Texas Cardiac arrhythmia Institute, St. David's Hospital, Austin, Texas